CLINICAL TRIAL: NCT06602232
Title: A Pilot, Safety and Clinical Activity, Phase 1b Study of DR-01 in Adults With Alopecia Areata or Vitiligo
Brief Title: A Study of DR-01 in Subjects With Alopecia Areata and Vitiligo
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dren Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DR-01-AIM-001
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-10

CONDITIONS: Alopecia Areata; Vitiligo
Keywords: AA; VT; Alopecia Areata; Alopecia; Vitiligo; Hair Diseases; Skin Diseases
MeSH Terms: conditions — Alopecia Areata; Vitiligo; Alopecia; Hair Diseases; Skin Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- DL1 of DR-01 (Experimental): Subjects in this arm will receive up to 6 months of dosing with DR-01 at dose level 1
  Interventions: Drug: DR-01
- DL2 of DR-01 (Experimental): Subjects in this arm will receive up to 6 months of dosing with DR-01 at dose level 2
  Interventions: Drug: DR-01
- DL3 of DR-01 (Experimental): Subjects in this arm will receive up to 6 months of dosing with DR-01 at dose level 3
  Interventions: Drug: DR-01
- DL4 of DR-01 (Experimental): Subjects in this arm will receive up to 6 months of dosing with DR-01 at dose level 4
  Interventions: Drug: DR-01

INTERVENTIONS:
Drug: DR-01 — DR-01 will be administered via IV infusion.

SUMMARY:
This is a multi-center, parallel-group, open-label, randomized, Phase 1b study to explore the safety, clinical activity, pharmacokinetics and pharmacodynamics of DR-01 in adults with Alopecia Areata or Vitiligo.

ELIGIBILITY:
General Inclusion Criteria

1. Subjects aged ≥ 18 with the ability to understand and comply with protocol-required study procedures, and voluntarily sign a written informed consent document.
2. Women of childbearing potential (postmenarcheal, has an intact uterus and at least 1 ovary, and is < 1 year postmenopausal) must agree to use a highly effective method of contraception (as specified in Section 13.1.1 or as permitted by regional regulatory authorities) from enrollment through at least 20 weeks after last dose of DR-01.
3. Male subjects must agree to use acceptable effective method(s) of contraception (as specified in Section 13.1.1 or as permitted by regional regulatory authorities) from enrollment through at least 20 weeks after last dose of DR-01.

   Alopecia Areata-Specific Inclusion Criteria
4. Diagnosed with moderate to severe AA with > 20% scalp hair loss at screening, according to SALT (Olsen 1999).
5. Current episode of AA lasting from > 6 months to < 10 years prior to screening.
6. No spontaneous improvement in the 6 months prior to screening or between screening and baseline (decrease in SALT score of ≤ 10, > 10 would be an improvement).
7. Patients with a current episode of AA lasting for ≥ 10 years may participate if there was regrowth in affected areas of the scalp over the 10 years prior to screening.
8. Agree not to use any AA treatments during the study (Exception: Chronic treatment with bimatoprost ophthalmic solution for eyelashes and chronic treatment with 5 alpha reductase inhibitors, oral or topical minoxidil).
9. Agree to not use adhesive wigs (other than banded perimeter wigs) during the study
10. Be willing to maintain the same hair style and hair dyeing throughout the study period.

    Subjects who shave their scalp must be willing to refrain from shaving their scalp for at least 2 weeks prior to each SALT assessment. Hair trimming outside the treatment areas to maintain the current hair style is permitted.

    Vitiligo-Specific Inclusion Criteria
11. Have active or stable non-segmental VT at screening and baseline defined as follows:

    1. Have a clinical diagnosis of non-segmental VT for at least 3 months; and
    2. Body surface area (BSA) involvement 4% to 60% excluding involvements at palms of the hands, dorsal aspect of fingers and thumbs including metacarpophalangeal joints, soles of the feet, or dorsal aspect of the feet; and
    3. BSA ≥ 0.25% involvement on the face excluding involvement at vermilion (confirmed by photographs at screening); and
    4. Subjects with active VT should have at least 1 active lesion defined as 1 of the following:

    i. New/extending lesion(s) in the past 3 months (confirmed by photographs or medical record); ii. Confetti-like lesion(s); iii. Trichrome lesion(s); iv. Koebner phenomenon/ phenomena (excluding Type 1 [history based isomorphic reaction]); e. Coexistence of halo nevus/nevi (also known as Sutton nevus/ nevi) is permitted.
12. If receiving concomitant medications for any reason other than VT, must be on a stable regimen, which is defined as not starting a new drug or changing dosage within 7 days or 5 half-lives (whichever is longer) prior to Day 1. Subject must be willing to stay on a stable regimen during the duration of the study.
13. Must agree to follow the usual and habitual exposure to sun light and not change the use of sunblock and not to use tanning booths, sun lamps or other ultraviolet light sources other than provided/requested by the study team during the study.

General Exclusion Criteria

Subjects meeting any of the following criteria are ineligible to participate in this study:

1. Participation in an investigational drug or device trial in which administration of an investigational drug or device occurred within 28 days or 5 half-lives of screening, whichever is shorter.
2. Use of live vaccines during the study and within 28 days prior to screening.
3. Known history of chronic alcohol abuse, IV drug abuse or illicit drug abuse within 1 year before screening.
4. Diagnosis or history of malignant disease within 5 years prior to baseline, with the exceptions of basal cell or squamous epithelial carcinomas of the skin that have been resected or cervical carcinoma in situ, with no evidence of recurrence within the 5 years prior to baseline.
5. Have had any surgical procedure (except for minor surgery requiring local or no anesthesia and without any complications or sequelae) within 12 weeks prior to screening, or any planned surgical procedure scheduled to occur during the study.
6. Any of the following types of infection within 28 days of screening or before randomization:

   1. Serious (requiring hospitalization, and/or IV anti-infective treatment).
   2. Chronic (duration of symptoms, signs, and/or treatment of 6 weeks or longer).
   3. Viral reactivation of CMV, EBV, VZV or HSV infection requiring systemic therapy in the last 2 years. Periodic HSV viral reactivation (e.g., cold sore) treated with a short course of systemic antiviral therapy within the last 2 years would not be exclusionary.
7. Any of the following:

   1. HIV infection.
   2. Current infection with HBV (i.e., positive for hepatitis B surface antigen and/or polymerase chain reaction positive for HBV DNA).
   3. Current infection with HCV (i.e., positive for HCV RNA).
8. Concurrent diagnosis or history of any autoimmune diseases other than AA or VT requiring systemic or topical immunotherapy.
9. Use of topical and oral JAK inhibitors within 4 and 8 weeks of randomization, respectively.
10. Use of lymphocyte depleting agents (e.g., rituximab, ocrelizumab, ofatumumab, ublituximab, thymoglobulin, alemtuzumab, etc.) within 6 months of screening or until lymphocyte counts have normalized.
11. Use of other biologics within 4 weeks of screening.
12. Use of oral immune suppressants (e.g., cyclosporine A, azathioprine, methotrexate, sulfasalazine, systemic corticosteroids, mycophenolate-mofetil,) within 28 days of screening. Topical steroid use is prohibited within 2 weeks of screening in VT and on scalp, eyebrows and eyelids in AA.
13. Intralesional steroid injection within 8 weeks of screening or within 5 half-lives, whichever is longer.
14. Herbal medications, including traditional Chinese medicine formulations, with unknown properties or known beneficial effects for VT or alopecia.
15. Untreated latent tuberculosis infection as indicated by IFNγ release assay, (appropriate therapy as defined by the World Health Organization and/or the United States Centers for Disease Control and Prevention). Without documentation of appropriate treatment.
16. Women who are currently pregnant or breastfeeding, or who intend to become pregnant or to breastfeed at any time during the study or within 20 weeks after receiving the last dose of DR-01.
17. Any other reason that may make the patient unsuitable for study participation, in the opinion of the Investigator or Medical Monitor
18. Subjects with intolerance or allergy to the investigational product or any of its components.
19. Estimated glomerular filtration rate < 30 mL/min/1.73m2 (using the Chronic Kidney Disease Epidemiology Collaboration formula (Levey 2009).
20. Total bilirubin >1.5 × upper limit of normal (ULN; > 3 × ULN if known Gilbert's disease).
21. Aspartate aminotransferase and alanine aminotransferase > 2.5 × ULN.

    Alopecia Areata-Specific Exclusion Criteria
22. Diffuse AA, other forms of alopecia and other active inflammatory diseases of the scalp.
23. Use of phototherapy, platelet-rich plasma injections or non-steroid topical immunosuppressives during the trial and within 12 weeks or 5 half-lives prior to screening.
24. Any history of disseminated/complicated herpes zoster.
25. Have a history of eczema herpeticum within 12 months prior to screening or a history of 2 or more episodes of eczema herpeticum in the past.

    Vitiligo-Specific Exclusion Criteria
26. Subjects that have other types of VT (including but not limited to segmental VT). Note: Mixed VT is permitted.
27. Currently have active forms of other hypopigmentation (including but not limited to Vogt-Koyanagi-Harada disease, malignancy-induced hypopigmentation [melanoma and mycosis fungoides], post-inflammatory hypopigmentation, pityriasis alba [minor manifestation of atopic dermatitis], senile leukoderma [age-related depigmentation], chemical/drug-induced leukoderma, ataxia telangiectasia, tuberous sclerosis, melasma, and congenital hypopigmentation disorders including piebaldism, Waardenburg syndrome, hypomelanosis of Ito, incontinentia pigmenti, dyschromatosis symmetrica hereditaria, xeroderma pigmentosum, and nevus depigmentosus). Note: Coexistence of halo nevus/nevi (also known as Sutton nevus/nevi) is permitted.
28. Currently have active forms of inflammatory skin disease(s) or evidence of skin conditions (including but not limited to morphea, discoid lupus, leprosy, syphilis, psoriasis, seborrheic dermatitis) at screening that in the opinion of the Investigator would interfere with evaluation of VT or response to treatment.
29. Use of permanent depigmentation treatment for VT and/or other types of pigmentation disorders (e.g., monobenzone or phenol) at any time.
30. Use of ultraviolet B phototherapy, psoralen ultraviolet A therapy, or other phototherapy within 4 weeks of screening.
31. Any history of disseminated/complicated or relapsing herpes zoster.
32. Have a history of eczema herpeticum within 12 months prior to screening or a history of 2 or more episodes of eczema herpeticum in the past.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events as assessed by CTCAE v5.0.(Safety and Tolerability) | Up to 12 months
Mean change from baseline in SALT score | At week 24
Mean change from baseline in VASI measures | At week 24

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rothenberg, MD, PhD, Study Director — Dren Bio
Locations (20):
- United States (12):
  - Dren Investigational Site, Northridge, California
  - Dren Investigational Site, Miami, Florida
  - Dren Investigational Site, Evans, Georgia
  - Dren Investigational Site, Meridian, Idaho
  - Dren Investigational Site, Indianapolis, Indiana
  - Dren Investigational Site, West Lafayette, Indiana
  - Dren Investigational Site, Worcester, Massachusetts
  - Dren Investigational Site, Troy, Michigan
  - Dren Investigational Site, Philadelphia, Pennsylvania
  - Dren Investigational Site, Pittsburgh, Pennsylvania
  - Dren Investigational Site, Chattanooga, Tennessee
  - Dren Investigational Site, San Antonio, Texas
- Australia (5):
  - Dren Investigational Site, Charlestown, New South Wales
  - Dren Investigational Site, Darlinghurst, New South Wales
  - Dren Investigational Site, Coorparoo, Queensland
  - Dren Investigational Site, South Yarra, Victoria
  - Dren Investigational Site, Fremantle, Washington
- New Zealand (3):
  - Dren Investigational Site, Auckland
  - Dren Investigational Site, Christchurch
  - Dren Investigational Site, Grafton

IPD SHARING:
Plan to Share IPD: No